CLINICAL TRIAL: NCT00003865
Title: Phase II Study of Two Dose Levels of Toremifene in the Treatment of Chemotherapy-Resistant Papillary Carcinoma of the Ovary
Brief Title: Toremifene in Treating Patients With Ovarian Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWCC-7096; CDR0000067029 (Registry Identifier: PDQ (Physician Data Query)); NCI-V99-1540
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer; ovarian serous cystadenocarcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Toremifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Toremifene (Experimental): All enrolled patients
  Interventions: Drug: toremifene

INTERVENTIONS:
Drug: toremifene

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of ovarian cancer cells. Hormone therapy using toremifene may fight ovarian cancer by reducing the production of estrogen.

PURPOSE: Randomized phase II trial to study the effectiveness of toremifene in treating patients who have recurrent or refractory ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effects of toremifene in terms of response rate, duration of response, duration of survival, and toxicity in patients with chemotherapy resistant papillary carcinoma of the ovary.
* Assess whether a dose response effect is likely for this regimen in these patients.
* Assess quality of life of these patients.

OUTLINE: This is a randomized study.

Patients receive one of two doses of oral toremifene daily for 4 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed before therapy and then every 4 weeks during therapy.

Patients are followed every 12 weeks until death.

PROJECTED ACCRUAL: The study was closed before any patient accrual.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed serous papillary carcinoma of the ovary

  * Recurrent or refractory disease following at least one regimen including paclitaxel, cisplatin, or carboplatin
* Measurable disease outside of irradiated field
* No CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* At least 16 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,800/mm^3
* Platelet count at least 125,000/mm^3
* No history of thrombosis or thromboembolic events

Hepatic:

* Bilirubin no greater than 2.0 mg/dL

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study
* No other concurrent second malignancy or prior malignancy within past 5 years, except basal or squamous cell skin cancer or curatively treated stage I carcinoma of the cervix
* No concurrent infection
* At least 3 days since prior fever (unless due to tumor)
* No other concurrent severe medical illness
* No HIV positivity

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No concurrent chemotherapy

Endocrine therapy:

* No prior tamoxifen or antiestrogen therapy

Radiotherapy:

* See Disease Characteristics
* At least 6 months since prior radiotherapy
* No concurrent radiotherapy except to symptomatic or potentially disabling bone lesion accompanied by other measurable disease

Surgery:

* Not specified

Other:

* No concurrent anticoagulants
* No other concurrent therapeutic trials

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-07-22 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Ahlgren, MD, Study Chair — George Washington University
Locations (1):
- George Washington University Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No